CLINICAL TRIAL: NCT04528446
Title: The Impact of Glomerular Disorders on Bone Quality and Strength
Acronym: BoneGN
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Thomas Nickolas, MD MS, Professor of Medicine, Columbia University
Other Study IDs: AAAS0922; R01DK119266 (NIH)
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Glomerular Disease; Bone Diseases, Metabolic; Bone Fracture
Keywords: Kidney Disease; Bone Fracture
MeSH Terms: conditions — Bone Diseases, Metabolic; Fractures, Bone; Kidney Diseases | interventions — Absorptiometry, Photon; Bone Density; Blood Specimen Collection; Urine Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — * Blood specimens (up to 50 ml or 3 ml/kg whichever is less) will be collected by venipuncture by a trained phlebotomist, and aliquots of serum and plasma will be stored at each visit for assays anticipated to be performed in one or two batches at the end of the study and biobanking for future studies.
  * Participants will be asked to provide 20 ml urine sample for biobanking at the time of the baseline and 12 month follow-up visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BoneGN participants: Participants who have already been recruited into the CureGN study, or meet its criteria.
  Interventions: Radiation: Dual-energy X-ray absorptiometry; Radiation: High Resolution Peripheral Quantitative Computed Tomography (HR-pQCT); Other: Blood draw and Urine collection; Other: Questionnaires

INTERVENTIONS:
Radiation: Dual-energy X-ray absorptiometry — DXA whole body, hip, spine, and radius at baseline, and 12-month visit.
  Other Names: Bone density
Radiation: High Resolution Peripheral Quantitative Computed Tomography (HR-pQCT) — HR-pQCT of the radius and tibia at baseline, and 12-month visit.
  Other Names: HR-pQCT
Other: Blood draw and Urine collection — The blood draw can be completed +/- 3 weeks from baseline or 12-month visit.
Other: Questionnaires — Questionnaires regarding fracture history, physical activity and dietary intake at baseline, and 12-month visit.

SUMMARY:
The primary objectives of this study are to: (1) determine the impact of glomerular disease on bone strength and (2) investigate the pathophysiologic underpinnings of impaired bone strength in glomerular disease.

DETAILED DESCRIPTION:
Children and adults with glomerular disease have unique and potentially modifiable risk factors for compromised bone health, but our current understanding of skeletal fragility in glomerular disease is lacking. In the first large population-based cohort study, we recently found that primary glomerular disease was independently associated with an increased risk of incident fracture, and that hip fracture risk was >2-fold greater in patients younger vs. older than 40 years of age. Mechanisms that drive increased fracture risk in glomerular disease are not clear but likely multifactorial. Our prior work demonstrated that glomerular disease is associated with disturbances in vitamin D and mineral metabolism, in addition to and exacerbated by reduced kidney function.

Patients with glomerular disease are also exposed to medications which may negatively impact bone health, most notably high-dose and long-term glucocorticoid therapy. Identifying modifiable factors that compromise bone strength will facilitate the development of strategies to reduce fractures and other skeletal complications across the life course. The proposed multi-center study will leverage the infrastructure of the NIH-funded Cure Glomerulopathy (CureGN) prospective cohort study and the resources of two health systems with expertise in state-of-the-art high-resolution bone imaging methods, to conduct the first prospective, longitudinal study to assess determinants of impaired bone quality and strength in glomerular disease.

ELIGIBILITY:
Inclusion Criteria for participants with glomerular disease:

1. CureGN participant or CureGN Eligible

   CureGN eligible is defined as having a diagnosis of Glomerulonephropathy (GN). Patients would otherwise be enrolled in be in CureGN study, except for lacking a minor entry criteria, such as:
   1. First diagnostic kidney biopsy within 5 years of CureGN study enrollment
   2. Access to first kidney biopsy report and/or slides or not being interested in study participation.
2. Males or females 5 to 55 years (premenopausal for women)
3. Females must have a negative urine/serum pregnancy test
4. Stable doses of nutritional vitamin D or active vitamin D therapy for at least 3 months before enrollment ((if on either form of Vitamin D)
5. Consent/Parental/guardian permission (informed consent) and if appropriate, child assent

Exclusion Criteria for all participants

1. Chronic Dialysis
2. Solid organ transplantation
3. Lower extremity amputations or non-ambulatory
4. Malignancy requiring chemotherapy or metastatic to bone
5. Metabolic bone disease (e.g., Paget's disease, primary hyperparathyroidism)
6. Endocrinopathy (current hyperthyroidism or untreated hypothyroidism, Cushing's syndrome)
7. Medical diseases (end stage liver disease, heart or lung disease, intestinal malabsorption)
8. Those treated with bisphosphonates, teriparatide, calcitonin, selective estrogen receptor modulators, estrogen, or phenytoin in the past 12 months
9. Previous bilateral wrist and tibia fractures
10. Pregnant or lactating females
11. Parents/guardians or participants who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Prospective cohort study of 150 CureGN participants (100 adults/50 children) will be evaluated at baseline and 12 months.
  The CureGN DCC at Arbor Research will identify CureGN participants eligible for inclusion. Recruitment of healthy participants will also occur by leveraging the services of the CHOP Recruitment Enhancement Core (REC), Pediatric Research Consortium (PeRC) and the RecruitMe tool provided by the Clinical Trials Office at CUMC. Healthy adult controls will be recruited from patients who receive outpatient care within the Penn Primary Care Networks, Penn employees and students, an extensive database of individuals who have participated in prior research studies at Penn and through local advertising on the Penn campus.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2019-06-14 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change in radius bone strength (failure load) | Baseline and 12 months
  HR-pQCT will be used to assess bone microarchitecture and generate micro-finite element analysis (µFEA)-based estimates of bone strength.
Change in tibia bone strength (failure load) | Baseline and 12 months
  HR-pQCT will be used to assess bone microarchitecture and generate micro-finite element analysis (µFEA)-based estimates of bone strength.

SECONDARY OUTCOMES:
Radius mid-shaft failure load | Up to 12 months
  Measured with HR-pQCT
Tibia mid-shaft failure load | Up to 12 months
  Measured with HR-pQCT
Cortical density of radius | Up to 12 months
  Measured with HR-pQCT
Cortical density of tibia | Up to 12 months
  Measured with HR-pQCT
Cortical thickness of radius | Up to 12 months
  Measured with HR-pQCT
Cortical thickness of tibia | Up to 12 months
  Measured with HR-pQCT
Areal bone mineral density (aBMD) at the hip | Up to 12 months
  Hip (total and femoral neck) is measured with dual-energy x-ray absorptiometry (DXA)
aBMD at forearm | Up to 12 months
  Forearm (one-third and ultradistal radius) is measured with DXA
aBMD at lumbar spine | Up to 12 months
  Lumbar spine is measured with DXA
Bone mineral content at the hip | Up to 12 months
  Hip (total and femoral neck) is measured with dual-energy x-ray absorptiometry (DXA)
Bone mineral content at forearm | Up to 12 months
  Forearm (one-third and ultradistal radius) is measured with DXA
Bone mineral content at lumbar spine | Up to 12 months
  Lumbar spine is measured with DXA

CONTACTS AND LOCATIONS:
Overall Officials: Thomas L. Nickolas, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Only investigators and study team members that have completed appropriate institutional review board (IRB) training/approval are eligible to collect and work on information collected from this study.

REFERENCES:
- [Background] Webster AC, Nagler EV, Morton RL, Masson P. Chronic Kidney Disease. Lancet. 2017 Mar 25;389(10075):1238-1252. doi: 10.1016/S0140-6736(16)32064-5. Epub 2016 Nov 23. PMID 27887750
- [Background] Floege J, Amann K. Primary glomerulonephritides. Lancet. 2016 May 14;387(10032):2036-48. doi: 10.1016/S0140-6736(16)00272-5. Epub 2016 Feb 25. PMID 26921911
- [Background] Saran R, Robinson B, Abbott KC, Agodoa LY, Albertus P, Ayanian J, Balkrishnan R, Bragg-Gresham J, Cao J, Chen JL, Cope E, Dharmarajan S, Dietrich X, Eckard A, Eggers PW, Gaber C, Gillen D, Gipson D, Gu H, Hailpern SM, Hall YN, Han Y, He K, Hebert H, Helmuth M, Herman W, Heung M, Hutton D, Jacobsen SJ, Ji N, Jin Y, Kalantar-Zadeh K, Kapke A, Katz R, Kovesdy CP, Kurtz V, Lavalee D, Li Y, Lu Y, McCullough K, Molnar MZ, Montez-Rath M, Morgenstern H, Mu Q, Mukhopadhyay P, Nallamothu B, Nguyen DV, Norris KC, O'Hare AM, Obi Y, Pearson J, Pisoni R, Plattner B, Port FK, Potukuchi P, Rao P, Ratkowiak K, Ravel V, Ray D, Rhee CM, Schaubel DE, Selewski DT, Shaw S, Shi J, Shieu M, Sim JJ, Song P, Soohoo M, Steffick D, Streja E, Tamura MK, Tentori F, Tilea A, Tong L, Turf M, Wang D, Wang M, Woodside K, Wyncott A, Xin X, Zang W, Zepel L, Zhang S, Zho H, Hirth RA, Shahinian V. US Renal Data System 2016 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2017 Mar;69(3 Suppl 1):A7-A8. doi: 10.1053/j.ajkd.2016.12.004. No abstract available. PMID 28236831
- [Background] Clark SL, Denburg MR, Furth SL. Physical activity and screen time in adolescents in the chronic kidney disease in children (CKiD) cohort. Pediatr Nephrol. 2016 May;31(5):801-8. doi: 10.1007/s00467-015-3287-z. Epub 2015 Dec 18. PMID 26684326
- [Background] Denburg MR, Kumar J, Jemielita T, Brooks ER, Skversky A, Portale AA, Salusky IB, Warady BA, Furth SL, Leonard MB. Fracture Burden and Risk Factors in Childhood CKD: Results from the CKiD Cohort Study. J Am Soc Nephrol. 2016 Feb;27(2):543-50. doi: 10.1681/ASN.2015020152. Epub 2015 Jul 2. PMID 26139439
- [Background] Phan V, Blydt-Hansen T, Feber J, Alos N, Arora S, Atkinson S, Bell L, Clarson C, Couch R, Cummings EA, Filler G, Grant RM, Grimmer J, Hebert D, Lentle B, Ma J, Matzinger M, Midgley J, Pinsk M, Rodd C, Shenouda N, Stein R, Stephure D, Taback S, Williams K, Rauch F, Siminoski K, Ward LM; Canadian STOPP Consortium. Skeletal findings in the first 12 months following initiation of glucocorticoid therapy for pediatric nephrotic syndrome. Osteoporos Int. 2014 Feb;25(2):627-37. doi: 10.1007/s00198-013-2466-7. Epub 2013 Aug 16. PMID 23948876
- [Background] Alem AM, Sherrard DJ, Gillen DL, Weiss NS, Beresford SA, Heckbert SR, Wong C, Stehman-Breen C. Increased risk of hip fracture among patients with end-stage renal disease. Kidney Int. 2000 Jul;58(1):396-9. doi: 10.1046/j.1523-1755.2000.00178.x. PMID 10886587